CLINICAL TRIAL: NCT02828670
Title: Role of T Follicular Helper Cells in Autoimmune Hemolytic Anemia (TFH in AIHA)
Acronym: TFH and AIHA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: AUDIA APJ 2014
Record Dates: First submitted 2016-06-23; First posted 2016-07-11 (Estimated); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- patient
  Interventions: Biological: blood sample; Procedure: spleen sample
- control
  Interventions: Biological: blood sample; Procedure: spleen sample

INTERVENTIONS:
Biological: blood sample
Procedure: spleen sample

SUMMARY:
T follicular helper (TFH) cells represent a T cell subset dedicated to the activation of B cells. They have been involved in the pathogenesis of autoimmune diseases in humans such as lupus and Sjögren disease. We recently showed that TFH are implicated in the activation of autoreactive B lymphocytes during ITP. Autoimmune hemolytic anemia (AIHA) is an autoimmune disease due to antibodies targeting red blood cells. To date, the role of TFH in the pathogenesis of AIHA is not known.

We hypothesize that AIHA is associated with an increase in the number and/or function of TFH, that could participate in the activation of autoreactive B lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of warm AIHA defined by

  * Hemoglobin <11 g/dl
  * Low haptoglobin level
  * Positive direct antiglobulin test (IgG or IgG + complement)
  * Reticulocyte count >120 G/L
* Patients

  * naive to treatment for hemolytic anemia or a in relapse
  * Older than 18 years
  * Able to understand written and spoken French
* Persons who have provided written consent

Control population

* Patients who have given consent
* Patients over 18 years
* Patients with cold agglutinin disease (progressive AIHA and different treatments of warm autoantibody AIHA) can be included as a sub-group of controls
* Patients with non-auto-immune hemolytic anemia (constitutional of enzymatic origin, membrane-related,…) can be included as a sub-group of controls

Exclusion Criteria:

* Patients without national health insurance
* Pregnancy or breast-feeding women
* Adults under guardianship
* Patients with cancer or malignant hemopathy
* Patients with an on-going infection
* Patients treated with corticoids or immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of warm AIHA Patients with non-auto-immune hemolytic anemia
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
the proportion of circulating T follicular helper lymphocytes (TFH) in patients with Autoimmune Hemolytic Anemia (AIHA) and in control subjects. | baseline
the proportion of circulating TFH in patients with Autoimmune Hemolytic Anemia (AIHA), at diagnosis and after 3 months of treatment with steroids | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France